CLINICAL TRIAL: NCT02340338
Title: Phase 1 Clinical Trial of the BioMed rTSST-1 Variant Vaccine in Healthy Adults
Brief Title: rTSST-1 Variant Vaccine Phase 1 First-in-man Trail
Acronym: rTSST-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedizinische Forschungs gmbH (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BioMed0713
Record Dates: First submitted 2014-11-21; First posted 2015-01-16 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Toxic Shock Syndrome; Vaccination; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Dose Group 1 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 100 ng
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 2 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 300 ng
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 3 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 1 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 4 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 3 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 5 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 10 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 6 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 30 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 0 (Placebo Comparator): Control: Al(OH)3 Adjuvant
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine

INTERVENTIONS:
Biological: rTSST-1 Variant Candidate Vaccine — In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.

SUMMARY:
Toxic Shock Syndrome (TSS) a severe condition with high morbidity and mortality results from the hosts overwhelming inflammatory response and cytokine storm. Staphylococcal superantigen toxins are the main causative agents. Toxic shock syndrome toxin (TSST-1) being responsible for almost all of menstruation associated and more than 50% of all other cases. There is no specific therapy.

The aim of this study is to demonstrate the safety and tolerability of the BioMed recombinant toxic shock syndrome toxin (rTSST-1) Variant Vaccine in healthy adults. The second aim of the study is to measure antibodies in the blood of these healthy volunteers which have been produced in response to treatment with the BioMed rTSST-1 Variant Vaccine. These antibodies are expected to be important in resistance against the diseases. 46 healthy adults, male and female, age 18-64 years will be assigned to 6 dose groups of the vaccine at the Department of Clinical Pharmacology of the Medical University of Vienna. The patients will be monitored for vital signs, hematology, clinical chemistry, blood cytokine level and antibodies against TSST-1. Immunization will be repeated 4 weeks after the first with the same dose.

DETAILED DESCRIPTION:
The BioMed rTSST-1 Variant Vaccine has been developed by Biomedizinische ForschungsgmbH as one component of a polyvalent staphylococcal vaccine for the prevention of toxic shock and hyperimmunization of donors for the production of TSST-1 immunoglobulin.

This is a prospective, partly randomized, parallel control, dose escalation study of the safety and immunogenicity of the BioMed rTSST1 Variant Vaccine compared to adjuvant in healthy adults.

28 - 3 days prior to entry into the study, 50 male and female subjects 18 - 64 years in age will be screened for eligibility , screening criteria to include physical examination, medical history, pregnancy/ adequate contraception in females, HIV Ab, hepatitis C virus antibodies (HCV Ab), hepatitis B antigen (HBs Ag) and TSST-1 Ab. 46 of these subjects will be entered into the study.

In a first step, two subjects will receive the adjuvanted Vaccine containing 100 ng rTSST-1 Ag and one subject will receive the adjuvant containing 0.2 mg Al(0H)3 only (Group 1). The subjects will be seen four times after immunization in a period of 14 days (6 h, 48 h + 2 hrs, 7 + 1 days and 14 + 2 days).Tests and examinations will include vital signs, hematology and clinical chemistry parameters, C-reactive protein, cytokines, TSST-Ab , local reactions and adverse events.

In the absence of clinically relevant adverse events , another three subjects will be entered into the study one week later, two of them to receive the adjuvanted Vaccine containing 300 ng rTSST-1 Ag, one receiving the adjuvant containing 0.6 mg Al(0H)3 (Group 2) and be followed for a period of 14 days as described above.

In the absence of clinically relevant adverse events , four more subjects will be entered into the study one week thereafter, three of them to receive the adjuvanted Vaccine containing 1 µg rTSST-1 Ag , one to receive adjuvant containing 1 mg Al(0H)3 alone (Group 3), and be followed for a period of 14 days in the manner described above.

Immunization will be repeated at the same dose level in each group one to two months after the first. Follow-up will be the same.

If immunogenicity can be shown after the second administration of the Vaccine containing 1 µg of rTSST-1 Ag, doses and sample sizes will be increased to Vaccine containing 3 µg , 10 µg, and 30 µg and adjuvant containing 1 mg Al(0H)3 in nine and three subjects in Groups 4 - 6, respectively. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level.

Subjects in Groups 4 - 6 will receive a second immunization at the respective dose level one to two months after the first, follow-up being the same as in Groups 1 - 3.

If there is no immune response in any dose group after the second immunization, a third injection will be given 4 - 8 weeks thereafter in dose groups of 1 µg (Groups 3 - 6) and above.

Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer.

Subjects to receive vaccine containing 3 µg rTSST-1 Ag or more will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* 18 - 64 years
* written informed consent
* physical exam: no abnormal findings unless considered irrelevant by the investigator
* uneventful medical history
* females: adequate contraception

Exclusion Criteria:

* pregnancy
* positive virology markers
* signs and symptoms of relevant autoimmunity
* TSST-1 Ab titer > 1:2000

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Eibl, MD, Study Director — Biomedizinische ForschungsgmbH; Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwameis M, Roppenser B, Firbas C, Gruener CS, Model N, Stich N, Roetzer A, Buchtele N, Jilma B, Eibl MM. Safety, tolerability, and immunogenicity of a recombinant toxic shock syndrome toxin (rTSST)-1 variant vaccine: a randomised, double-blind, adjuvant-controlled, dose escalation first-in-man trial. Lancet Infect Dis. 2016 Sep;16(9):1036-1044. doi: 10.1016/S1473-3099(16)30115-3. Epub 2016 Jun 10. PMID 27296693

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Group 1: Treatment: rTSST-1 Variant Candidate Vaccine 100 ng
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 2: Treatment: rTSST-1 Variant Candidate Vaccine 300 ng
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 3: Treatment: rTSST-1 Variant Candidate Vaccine 1 µg
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 4: Treatment: rTSST-1 Variant Candidate Vaccine 3 µg
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 5: Treatment: rTSST-1 Variant Candidate Vaccine 10 µg
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 6: Treatment: rTSST-1 Variant Candidate Vaccine 30 µg
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
- Dose Group 0: Control: Al(OH)3 Adjuvant
  rTSST-1 Variant Candidate Vaccine: In the absence of adverse events classified as clinically relevant, interval between dose escalations 1 week. Immunization to be repeated at the same dose level 1 - 2 months later. If immunogenicity can be shown after the second administration of 1 µg, the sample size will be increased from 3 + 1 to 9 + 3. Otherwise, the sample size of 3 + 1 will continue until immunogenicity is seen at a higher dose level. If there is no immune response in any dose group after the second immunization, a third injection will be given 4 -8 weeks thereafter in dose groups of 1 µg and above.
  Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer .
  Patients 3 µg or more will be randomized.
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 0
Started | 2 (2 vaccine + 1 placebo) | 2 (2 vaccine + 1 placebo) | 3 (3 vaccine + 1 placebo) | 9 (9 vaccine + 3 placebo) | 9 (9 vaccine + 3 placebo) | 9 (9 vaccine + 3 placebo) | 12 (Placebos were randomly assigned to dose groups 1-6, included in the 46 participants.)
Completed | 2 | 2 | 3 | 9 | 9 | 9 (1 withdrew voluntarily after the first immunization; safety and serum assessment completed.) | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 0 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 9 | 9 | 9 | 12 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 9 | 9 | 9 | 12 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (9.9) | 37.5 (13.4) | 36.3 (5.1) | 36.2 (10.9) | 33.7 (11.7) | 27.7 (7.2) | 34.4 (8.5) | 34.0 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4 | 6 | 7 | 6 | 27
  Male | 2 | 0 | 1 | 5 | 3 | 2 | 6 | 19
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 2 | 3 | 9 | 9 | 9 | 12 | 46
Safety and Immunogenicity assessment. [Number; unit: participants] — Initial screening of antibody titers of participants of all groups since high titers were among exclusion criteria. For this reason, all patients included were assessed for antibody titers at that time point.
  participants | 2 | 2 | 3 | 9 | 9 | 9 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Clinical observations and clinical laboratory values
Time Frame: through day 70
Measure: Number; unit: participants with any solicited AE
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 0
Number analyzed (Participants) | 2 | 2 | 3 | 9 | 9 | 9 | 12
participants with any solicited AE | 1 | 1 | 2 | 7 | 8 | 7 | 9

2. Secondary Outcome: Number of Participants With Seroconversion
Description: ELISA IgG against rTSST-1
Time Frame: through day 70
Measure: Number; unit: participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 0
Number analyzed (Participants) | 2 | 2 | 3 | 9 | 9 | 9 | 12
participants | 1 | 2 | 1 | 8 | 9 | 6 | 0

ADVERSE EVENTS:
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/9 | 0/9 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 2/3 | 7/9 | 8/9 | 7/9 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group 1 (N=2) | Dose Group 2 (N=2) | Dose Group 3 (N=3) | Dose Group 4 (N=9) | Dose Group 5 (N=9) | Dose Group 6 (N=9) | Dose Group 0 (N=12)
Mild to moderate reactions (General disorders) | 1 | 1 | 2 | 7 | 8 | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No